CLINICAL TRIAL: NCT00192634
Title: A Randomised, Open-label Trial to Assess the Safety and Efficacy of Switching to Tenofovir-emtricitabine or Abacavir-lamivudine: The STEAL Study.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Prof Sean Emery, The National Centre in HIV Epidemiology and Clinical Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEAL; ACTRN012605000505606
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: HIV Infections
Keywords: HIV; Antiretroviral therapy; nucleoside analogue reverse transcriptase; fixed dose combination; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; abacavir; Lamivudine; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Abacavir 600mg/Lamivudine 300mg
  Interventions: Drug: Abacavir 600mg - Lamivudine 300mg
- 2 (Active Comparator): Tenofovir 300mg/emtricitabine 200mg
  Interventions: Drug: Emtricitabine 200mg - Tenofovir 300mg

INTERVENTIONS:
Drug: Emtricitabine 200mg - Tenofovir 300mg — 1 tablet once daily for 96 weeks
  Other Names: Truvada
  Arms: 2
Drug: Abacavir 600mg - Lamivudine 300mg — 1 tablet once daily for 96 weeks
  Other Names: Kivexa
  Arms: 1

SUMMARY:
Combination antiretroviral therapy for the treatment of HIV has a high pill burden. Two dual-tablets, abacavir-lamivudine and tenofovir-emtricitabine, are now licensed in the United States and will be available in Australia in December 2005. Data available suggest that the potency of these tablets are similar in controlling replication of the HIV virus, but not have not been directly compared in regard to clinically significant toxicities. We therefore aim to compare the overall safety and efficacy of the two dual-tablets over a 2 year period in HIV infected adults. We hypothesise that the two dual-NRTI treatments will be similar in efficacy and safety.

DETAILED DESCRIPTION:
The aim of this study is to compare the overall safety and efficacy of two dual-NRTI, once daily, tablets over a 2 year period in HIV infected adults.

The study is a randomised, multi-centre, 2 year study of two dual NRTI, once daily tablets in subjects with HIV, currently taking two individual NRTIs as part of their therapy. 350 subjects will be randomised in a 1:1 ratio to either:

1. tenofovir (TDF) 300mg + emtricitabine (FTC) 200mg OR
2. abacavir (ABC) 600mg + lamivudine (3TC) 300mg. Subjects will cease their current individual NRTI treatment, commence their randomised dual NRTI tablet, and continue on their current NNRTI or PI therapy.

Subjects will be stratified by the type of NRTI they are currently taking (ABC, TDF or other); whether they are currently taking a protease inhibitor (yes or no); and by the site where they are randomised. A study plan is enclosed

Subjects will be closely monitored (at 1 month and then every 3 months until week 96) for safety by evaluating the incidence and severity of adverse effects/abnormal laboratory parameters. Study investigations enclosed. It is optional whether subjects also provide plasma, serum and cells (PBMCs) for storage. These samples will be available for analysis for sub-studies agreed to through the IVRN expression of interest network.

ELIGIBILITY:
Inclusion Criteria:

* documented HIV infection
* age at least 18 years
* stable (≥ to 12 weeks) ART including at least two NRTIs, currently well tolerated, with no plan to change any other component of the ART regimen at or after baseline
* HIV RNA < 50 copies/mL plasma for the preceding 12 weeks
* GFR ≥ 70 mL/min/1.73m2 (estimated by the abbreviated MDRD equation23 estimated GFR = 186 x ([SCR/88.4]-1.154) x age-0.203 x (0.742 if female) x (1.210 if African-American)
* provision of written, informed consent

Exclusion Criteria:

* HLA-B*5701 positive at screening OR evidence of previous ABC hypersensitivity OR clinical failure in participants taking abacavir for at least 30 days
* current therapy comprising triple NRTI therapy alone
* current use of ABC/3TC FDC (Kivexa) or TDF/FTC FDC (Truvada)
* history of non-traumatic osteoporotic fracture
* prior hypersensitivity or intolerance to ABC, 3TC, TDF or FTC
* prior clinical failure to a regimen containing ABC or TDF
* prior use of TDF for control of previously active hepatitis B (HBsAg+ or HBV DNA+) in patients likely to be resistant to 3TC/FTC
* current therapy including unboosted atazanavir
* concurrent use of aminoglycosides, IV amphotericin B, cidofovir, cisplatin, foscarnet, IV pentamidine, probenecid, adefovir or immunomodulatory agents
* clinical evidence of cirrhosis (e.g. smooth liver, no features of portal hypertension)
* creatinine clearance < 50 mL/min (estimated by the Cockcroft-Gault equation)18,19

  * Male: (140 - age in years) x (wt in kg) = CLCr (mL/min) 0.814 x (serum creatinine in µmol/L)
  * Female:(140 - age in years) x (wt in kg) x 0.85 = CLCr (mL/min) 0.814 x (serum creatinine in µmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2005-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
virological failure defined by HIV RNA>400copies/mL plasma on 2 consecutive occasions ³4 wks apart(Roche Amplicor v1.5, LLD 50 copies/mL) | Week 48

SECONDARY OUTCOMES:
plasma HIV RNA<50copies/mL; time to virological failure (VF); virological resistance in those with VF; all SAEs; use of concomitant meds for toxicity; adherence; QoL; CD4+lymphocyte count; full blood count; biochemistry; lipid parameters | Week 48 and 96
glycaemic parameters; DEXA parameters; resolution of AEs; progression to AIDS; death; discontinuation of ART. | Week 48 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Carr, MD FRACP FRCPA, Principal Investigator — Kirby Institute
Locations (31):
- Australia (31):
  - Holdsworth House General Practice - Byron Bay, Byron Bay, New South Wales
  - Lismore Sexual Health Clinic - Northen Rivers Area Health Service, Lismore, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - 407 Doctors, Sydney, New South Wales
  - Albion Street Centre, Sydney, New South Wales
  - Holdsworth House General Practice, Sydney, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - Taylor Square Private Clinic, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Clinic 16, Royal North Shore Hospital, Sydney, New South Wales
  - Burwood Road Practice, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Liverpool Health Service, Sydney, New South Wales
  - QLD Health - AIDS Medical Unit, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Gladstone Road Medical Centre, Brisbane, Queensland
  - Doll's House Clinic - Cairns Base Hospital, Cairns, Queensland
  - Gold Coast Sexual Health Clinic, Miami, Queensland
  - Clinic 87, Nambour Hospital, Nambour, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Care and Prevention Programme - Adelaide University, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Carlton Clinic, Melbourne, Victoria
  - Melbourne Sexual Health Centre, Melbourne, Victoria
  - Prahran Market Clinic, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - The Centre Clinic, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Royal Perth Hospital, Perth, Western Australia

REFERENCES:
- [Result] http://www.retroconference.org/AbstractSearch/Default.aspx?Conf=18
- [Result] Martin A, Bloch M, Amin J, Baker D, Cooper DA, Emery S, Carr A. Simplification of antiretroviral therapy with tenofovir-emtricitabine or abacavir-Lamivudine: a randomized, 96-week trial. Clin Infect Dis. 2009 Nov 15;49(10):1591-601. doi: 10.1086/644769. PMID 19842973
- [Derived] Haskelberg H, Pocock N, Amin J, Ebeling PR, Emery S, Carr A; STEAL study investigators; Allworth A. Hip structural parameters over 96 weeks in HIV-infected adults switching treatment to tenofovir-emtricitabine or abacavir-lamivudine. PLoS One. 2014 Apr 10;9(4):e94858. doi: 10.1371/journal.pone.0094858. eCollection 2014. PMID 24722774
- [Derived] Haskelberg H, Cordery DV, Amin J, Kelleher AD, Cooper DA, Emery S; STEAL Study Group. HLA alleles association with changes in bone mineral density in HIV-1-infected adults changing treatment to tenofovir-emtricitabine or abacavir-lamivudine. PLoS One. 2014 Mar 28;9(3):e93333. doi: 10.1371/journal.pone.0093333. eCollection 2014. PMID 24681993
- See also: National Centre in HIV Epidemiology and Clinical Research Homepage — http://www.med.unsw.edu.au/nchecr/